CLINICAL TRIAL: NCT02333578
Title: A Phase I/II Pilot Clinical Trial to Evaluate the Efficacy and Safety of Ebola Virus Disease (EVD) Convalescent Plasma (ECP) for Treatment of EVD
Brief Title: Clinical Trial to Evaluate the Efficacy and Safety of Convalescent Plasma for Ebola Treatment
Acronym: EVD001
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Clinical Research Management, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EVD001
Record Dates: First submitted 2015-01-05; First posted 2015-01-07 (Estimated); Last update posted 2015-01-07 (Estimated); Status verified 2015-01

CONDITIONS: Ebola Virus Disease
MeSH Terms: conditions — Hemorrhagic Fever, Ebola | interventions — COVID-19 Serotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Convalescent Plasma Treatment (Experimental): This pilot trial will treat subjects in the ECP Group with ECP derived from two donors. ECP will be provided as ECPSDU each comprising 90 - 110mL of plasma from two individual ABO-compatible donors. Two ECPSDU will be administered as immediately sequential infusions. Subjects may receive up to three doses of ECP not less than 48 hours apart. ECP will be provided as Plasma Frozen Within 24 Hours After Phlebotomy (PF24).
  Interventions: Procedure: Convalescent Plasma Treatment

INTERVENTIONS:
Procedure: Convalescent Plasma Treatment — This pilot trial will treat subjects in the ECP Group with ECP derived from two donors. ECP will be provided as ECPSDU each comprising 90 - 110mL of plasma from two individual ABO-compatible donors. Two ECPSDU will be administered as immediately sequential infusions. Subjects may receive up to three doses of ECP not less than 48 hours apart. ECP will be provided as Plasma Frozen Within 24 Hours After Phlebotomy (PF24).

SUMMARY:
A Phase I/II Pilot Clinical Trial to Evaluate the Efficacy and Safety of Ebola Virus Disease (EVD) Convalescent Plasma (ECP) for treatment of EVD.

DETAILED DESCRIPTION:
This pilot trial will treat subjects in the ECP Group with ECP derived from two donors. ECP will be provided as ECPSDU each comprising 90 - 110mL of plasma from two individual ABO-compatible donors. Two ECPSDU will be administered as immediately sequential infusions. Subjects may receive up to three doses of ECP not less than 48 hours apart. ECP will be provided as Plasma Frozen Within 24 Hours After Phlebotomy (PF24) as described in Section 6.1. Pre-treatment and frequent post-treatment blood specimens for assay of anti-EBOV antibody and EBOV viral load by RT-PCR will be obtained from subjects. The pharmacodynamic effect of ECP anti-EBOV, including neutralization titers, on viral load will be examined in the ECP Group. Changes of individual and treatment group clinical and laboratory parameters with time will be described. Between-group and within-group will examine interactions of clinical parameters, outcome, ECP total dose, EBOV viral load, and anti-EBOV (IgG ELISAs for Zaire GP residues 1-649 and irradiated Zaire virus, and anti-EBOV PRNT). The MEWS will be assessed as a prognostic tool in the Screened Control Group. Efficacy of ECP will be assessed primarily by comparison of survival to hospital discharge between the ECP Group and the Screened Control Group.

ELIGIBILITY:
Inclusion Criteria:

* Adult male or female 18 years of age or older
* Confirmed case of EVD (CDC case definitions 14 SEP 2014)
* Admission to the hospital no more than 48 hours prior to availability of investigational product
* Able and willing to provide informed consent or family member who is willing and able to provide informed consent if potential subject is unable to consent
* Venous access adequate for administration of plasma
* Females only: negative qualitative urine Beta-HCG test

Exclusion Criteria:

* Prior history of severe transfusion reaction
* Fluid overload or other condition that would contraindicate administration of plasma at the protocol- specified doses
* History of blood product transfusion within 30 days prior to enrollment
* Prior treatment with any other specific experimental anti-EVD product or expectation to receive another experimental anti-EVD product during the course of the study (does not include general supportive care or nutritional supplements routinely administered to all hospitalized patients with EVD)
* Unresponsive on AVPU (Alert, Voice Responsive, Pain Responsive, Unresponsive) testing

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2014-11; Primary Completion 2015-04 (Estimated); Study Completion 2015-06 (Estimated)

PRIMARY OUTCOMES:
EBOV viral load in blood of ECP Group as measured by quantitative FDA-authorized DoD EZ1 Real-time RT-PCR using USAMRIID research protocol | 12 Weeks

CONTACTS AND LOCATIONS:
Overall Officials: Jerry Brown, MD, Principal Investigator — ELWA Hospital
Locations (1):
- ELWA-2 Ebola Treatment Unit, Monrovia, Liberia

REFERENCES:
- [Derived] Brown JF, Dye JM, Tozay S, Jeh-Mulbah G, Wohl DA, Fischer WA 2nd, Cunningham CK, Rowe K, Zacharias P, van Hasselt J, Norwood DA, Thielman NM, Zak SE, Hoover DL. Anti-Ebola Virus Antibody Levels in Convalescent Plasma and Viral Load After Plasma Infusion in Patients With Ebola Virus Disease. J Infect Dis. 2018 Jul 13;218(4):555-562. doi: 10.1093/infdis/jiy199. PMID 29659889